CLINICAL TRIAL: NCT03834363
Title: Morphine or Fentanyl for Refractory Dyspnea in COPD
Acronym: MoreFoRCOPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huib A.M. Kerstjens (Other)
Collaborators: Dutch Foundation for Asthma Prevention (Unknown); Innovatiefonds Zorgverzekeraars (Other)
Responsible Party: Sponsor-Investigator, Huib A.M. Kerstjens, Full professor pulmonology, head of department pulmonology and tuberculosis, principal investigator., University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MoreFoRCOPD
Record Dates: First submitted 2019-01-11; First posted 2019-02-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: COPD
Keywords: COPD; Refractory Dyspnea; Morphine; Fentanyl
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Fentanyl; Morphine

STUDY DESIGN:
Intervention Model Description: Crossover, double blind, double dummy Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For both morphine retard capsules as fentanyl patches there is a placebo available. Participants will be treated in each period with both tablets and a patch. (morphine capsules+placebo patch, placebo capsules+fentanyl patch, placebo capsules+ placebo patch.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Morphine capsules and Placebo patch (Active Comparator): Morphine retard 10 mg twice daily Placebo patch, change every three days.
  Interventions: Drug: Morphine Retard; Drug: Placebo patch
- Placebo capsules and Fentanyl patch (Experimental): Placebo capsules twice daily Fentanyl patch 12 mcg/hr, change every three days
  Interventions: Drug: Fentanyl; Drug: Placebo oral capsule
- Placebo capsules and Placebo patch (Placebo Comparator): Placebo capsules twice daily Placebo patch, change every three days
  Interventions: Drug: Placebo patch; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Fentanyl — Fentanylpatch 12 mcg/hr, change patch every three days.
  Other Names: Fentanyl Matrix
  Arms: Placebo capsules and Fentanyl patch
Drug: Morphine Retard — Morphine retard capsules 10 mg bid.
  Other Names: Morphine
  Arms: Morphine capsules and Placebo patch
Drug: Placebo patch — Placebo patch, change patch every three days.
  Arms: Morphine capsules and Placebo patch; Placebo capsules and Placebo patch
Drug: Placebo oral capsule — Placebo oral capsule bid
  Arms: Placebo capsules and Fentanyl patch; Placebo capsules and Placebo patch

SUMMARY:
Rationale: The most important complaint in severe COPD is dyspnea which is associated with a diminished exercise tolerance, reduced quality of life and can lead to anxiety and depression. If dyspnea continues to exist despite optimal therapy it is called refractory dyspnea. There is evidence that morphine is effective and can safely be prescribed for treating refractory dyspnea.

However, a Dutch study recently showed that few pulmonologists actually prescribe opioids for this indication. The main reasons for this are concerns about side effects and respiratory insufficiency as well as negative emotions for the patient and families at the thought of using morphine.

Most studies investigating opioids for treatment of dyspnea are conducted with morphine tablets, and only a part of these patients suffered from COPD. To our knowledge there has not been a randomized controlled trial investigating fentanyl patches for refractory dyspnea in COPD patients. However, studies comparing fentanyl and morphine in pain management show that patients may prefer fentanyl patches and have less problems with obstipation.

Objective: There are three main objectives for this study.

First, the investigators will investigate the following hypothesis: Both fentanyl and morphine provide a reduction of dyspnea which is better than placebo. Fentanyl has less side effects than morphine.

Secondly, with this Dutch multi-center study the investigators would like to enlarge the evidence base and contribute to the experience with opioids for refractory dyspnea in COPD thereby greatly facilitating its implementation in the Netherlands.

Finally, the investigators will develop and evaluate educational material about opioid use for dyspnea in COPD.

Study design: This is a multi-center double blind, double-dummy cross-over randomized placebo-controlled trial with three study arms. A total of 60 COPD patients will be included in this study.

Participants will be treated sequentially with three combinations of medication and/or placebo medication in a random order. They will receive either a Fentanyl patch in combination with placebo tablets, a placebo patch with Morphine Slow release tablets or a placebo patch with placebo tablets. Main study parameters/endpoints: The primary endpoint is change in dyspnea sensation Secondary endpoints are change in HR-QoL, anxiety, sleep quality, hypercapnia and the number and seriousness of side effect.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years.
* Read, understood and signed the Informed Consent form.
* COPD GOLD class III or IV, according to GOLD criteria (Post-bronchodilation FEV/FVC <70% and FEV1 < 50%pred.
* Complaints of refractory dyspnea as established by patient and doctor.
* mMRC score ≥ 3.
* Life expectancy of ≥ 2 months.
* Optimized standard therapy according to Dutch LAN guideline for diagnosis and treatment of COPD.

Exclusion Criteria:

* Other severe disease with chronic pain or chronic dyspnea (a non substantial component of left sided heart failure is acceptable).
* Current use of opioids for whatever indication.
* Allergy / intolerance for opioids
* Psychiatric disease, not related to severe COPD.
* Exacerbation of COPD 8 weeks prior to inclusion or between screening and randomization.
* Problematic (leading to medical help or social problems) substance abuse during the last five years.
* Active malignancy, with the exception of planocellular or basal cell carcinoma of the skin.
* eGFR <15 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Change in dyspnea sensation | Daily during the six week treatment period
  Change in dyspnea sensation measured on a Numeric Rating Scale from 0 to 10. A lower score represents a better outcome.

SECONDARY OUTCOMES:
Change in CCQ (HR-QoL) | Daily during the six week treatment period
  Change in HR-QoL measured with the Clinical COPD Questionnaire. Scores range from 0 to 6. Lower values represent a better outcome.
Change in CRQ (HR-QoL) | 4 times during the six week treatment period: baseline, 2 weeks, 4 weeks, 6 weeks.
  Change in HR-QoL measured with Chronic Respiratory Disease Questionnare. Scores range from 1 to 7. A higher score represents a better outcome.
Change in CRQ mastery (HR-QoL) | 4 times during the six week treatment period: baseline, 2 weeks, 4 weeks, 6 weeks.
  Change in HR-QoL measured with Chronic Respiratory Disease Questionnare, domain Mastery. Scores range from 1 to 7. A higher score represents a better outcome.
Change on the HADS-A questionnaire (Anxiety) | 4 times during the six week treatment period: baseline, 2 weeks, 4 weeks, 6 weeks.
  Change on the Hospital Anxiety and Depression Scale-anxiety subscale. Scores range from 0 to 21. A lower score represents a better outcome.
Side effects | Daily during the six week treatment period
  Reported spontaneously in a daily patient diary and specifically, both open and named side effects at planned visits.
Hypercapnia | 4 times during the six week treatment period: baseline, 2 weeks, 4 weeks, 6 weeks.
  Change in pCO2 in capillary blood gas analysis
Sleep quality | Daily during the six week treatment period
  Change on a Numeric Rating Scale from 0 to 10. A lower score represents a better outcome.
Continued opioid use | Once, three months after the end of the treatment period
  Asked three months after the end of the treatment period

OTHER OUTCOMES:
Survival | One week after the end of the treatment period, which is 7 weeks after start of the study.
  Measured one week after the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Huib AM Kerstjens, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (10):
- Netherlands (10):
  - Wilhelmina Ziekenhuis Assen, Assen, Drenthe
  - Elkerliek Ziekenhuis, Helmond, North Brabant
  - Noordwest Ziekenhuisgroep Alkmaar, Alkmaar, North Holland
  - Rode Kruis Ziekenhuis, Beverwijk, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala Klinieken, Zwolle, Overijssel
  - Ommelander Ziekenhuis Groningen, Scheemda, Provincie Groningen
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, ICF
Time Frame: After publication of results Unlimited
Access Criteria: Clear description of goals for asking

REFERENCES:
- [Background] Blinderman CD, Homel P, Billings JA, Tennstedt S, Portenoy RK. Symptom distress and quality of life in patients with advanced chronic obstructive pulmonary disease. J Pain Symptom Manage. 2009 Jul;38(1):115-23. doi: 10.1016/j.jpainsymman.2008.07.006. Epub 2009 Feb 20. PMID 19232893
- [Background] Wiseman R, Rowett D, Allcroft P, Abernethy A, Currow DC. Chronic refractory dyspnoea--evidence based management. Aust Fam Physician. 2013 Mar;42(3):137-40. PMID 23529525
- [Background] Abernethy AP, Currow DC, Frith P, Fazekas BS, McHugh A, Bui C. Randomised, double blind, placebo controlled crossover trial of sustained release morphine for the management of refractory dyspnoea. BMJ. 2003 Sep 6;327(7414):523-8. doi: 10.1136/bmj.327.7414.523. PMID 12958109
- [Background] Jennings AL, Davies AN, Higgins JP, Gibbs JS, Broadley KE. A systematic review of the use of opioids in the management of dyspnoea. Thorax. 2002 Nov;57(11):939-44. doi: 10.1136/thorax.57.11.939. PMID 12403875
- [Background] Janssen DJ, de Hosson SM, bij de Vaate E, Mooren KJ, Baas AA. Attitudes toward opioids for refractory dyspnea in COPD among Dutch chest physicians. Chron Respir Dis. 2015 May;12(2):85-92. doi: 10.1177/1479972315571926. Epub 2015 Feb 12. PMID 25676931
- [Background] Simon ST, Koskeroglu P, Gaertner J, Voltz R. Fentanyl for the relief of refractory breathlessness: a systematic review. J Pain Symptom Manage. 2013 Dec;46(6):874-86. doi: 10.1016/j.jpainsymman.2013.02.019. Epub 2013 Jun 4. PMID 23742735
- [Background] Payne R, Mathias SD, Pasta DJ, Wanke LA, Williams R, Mahmoud R. Quality of life and cancer pain: satisfaction and side effects with transdermal fentanyl versus oral morphine. J Clin Oncol. 1998 Apr;16(4):1588-93. doi: 10.1200/JCO.1998.16.4.1588. PMID 9552070
- [Background] Allan L, Hays H, Jensen NH, de Waroux BL, Bolt M, Donald R, Kalso E. Randomised crossover trial of transdermal fentanyl and sustained release oral morphine for treating chronic non-cancer pain. BMJ. 2001 May 12;322(7295):1154-8. doi: 10.1136/bmj.322.7295.1154. PMID 11348910
- [Background] Johnson MJ, Bland JM, Oxberry SG, Abernethy AP, Currow DC. Clinically important differences in the intensity of chronic refractory breathlessness. J Pain Symptom Manage. 2013 Dec;46(6):957-63. doi: 10.1016/j.jpainsymman.2013.01.011. Epub 2013 Apr 19. PMID 23608121
- [Background] Currow DC, McDonald C, Oaten S, Kenny B, Allcroft P, Frith P, Briffa M, Johnson MJ, Abernethy AP. Once-daily opioids for chronic dyspnea: a dose increment and pharmacovigilance study. J Pain Symptom Manage. 2011 Sep;42(3):388-99. doi: 10.1016/j.jpainsymman.2010.11.021. Epub 2011 Mar 31. PMID 21458217
- [Background] Jensen D, Alsuhail A, Viola R, Dudgeon DJ, Webb KA, O'Donnell DE. Inhaled fentanyl citrate improves exercise endurance during high-intensity constant work rate cycle exercise in chronic obstructive pulmonary disease. J Pain Symptom Manage. 2012 Apr;43(4):706-19. doi: 10.1016/j.jpainsymman.2011.05.007. Epub 2011 Dec 14. PMID 22168961
- [Background] Hui D, Kilgore K, Frisbee-Hume S, Park M, Liu D, Balachandran DD, Bruera E. Effect of Prophylactic Fentanyl Buccal Tablet on Episodic Exertional Dyspnea: A Pilot Double-Blind Randomized Controlled Trial. J Pain Symptom Manage. 2017 Dec;54(6):798-805. doi: 10.1016/j.jpainsymman.2017.08.001. Epub 2017 Aug 10. PMID 28803087
- [Derived] van Dijk M, Mooren KJM, van den Berg JK, van Beurden-Moeskops WJC, Heller-Baan R, de Hosson SM, Lam-Wong WY, Peters L, Pool K, Kerstjens HAM. Opioids in patients with COPD and refractory dyspnea: literature review and design of a multicenter double blind study of low dosed morphine and fentanyl (MoreFoRCOPD). BMC Pulm Med. 2021 Sep 10;21(1):289. doi: 10.1186/s12890-021-01647-8. PMID 34507574